CLINICAL TRIAL: NCT05357521
Title: Feasibility and Preliminary Data on the Interplay Between Oxytocin and Cortisol During Stress in Borderline Personality Disorder
Brief Title: Interplay Between Oxytocin and Cortisol During Stress in Borderline Personality Disorder
Acronym: OXT-CORT-BPD
Status: Completed | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Tatiana Aboulafia Brakha, PhD, University of Geneva, Switzerland
Other Study IDs: 2002-00067
Record Dates: First submitted 2022-03-05; First posted 2022-05-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-03

CONDITIONS: Borderline Personality Disorder; Oxytocin
Keywords: cortisol; tsst; borderline personnality; stress
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Borderline personality disorder: female patients between 18 and 25 years old meeting DSM V criteria for borderline personality disorder
  Interventions: Other: stress test
- Control: female participants between 18 and 25 years old, with no psychiatric history, not meeting criteria for borderline personality disorder
  Interventions: Other: stress test

INTERVENTIONS:
Other: stress test — TSST- psychosocial stress test

SUMMARY:
This study aims to determine the feasibility and preliminary data on the interaction between oxytocin and cortisol during stress in borderline personnality disorder.

DETAILED DESCRIPTION:
The investigators will recruit 50 female patients with borderline personnality disorder and 50 controls with no psychiatric diagnosis, aged between 18 and 25 years old.

salivary cortisol daily curve ( 6 measures during the day) will be measured in participant's naturalistic environnement, together with salivary oxytocin. In addition, salivary oxytocin and cortisol will be measured during a psychosocial stress task and recovery.

ELIGIBILITY:
Inclusion Criteria:

* Borderline personality disorder-DSM V

Exclusion Criteria:

* Schizophrenia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with and without borderline personality disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol | Baseline
  salivary cortisol measured with salivettes (swabs)
Salivary cortisol | Change in one day (circadian cortisol with 6 measures within one day
  salivary cortisol measured with salivettes (swabs)
Salivary cortisol | Change during experimental task (up to 2 hours)
  salivary cortisol measured with salivettes (swabs)
Salivary oxytocin | Baseline
  salivary oxytocin measured with salivettes (swabs)
Salivary oxytocin | Two measures within one day
  salivary oxytocin measured with salivettes (swabs)
Salivary oxytocin | Change during experimental task (up to 2 hours)
  salivary oxytocin measured with salivettes (swabs)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Aboulafia Brakha, PhD, Principal Investigator — Geneva Univeristy hospital
Locations (1):
- Young Adult Psychiatric Unit, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided